CLINICAL TRIAL: NCT00454909
Title: Study to Assess Immunogenicity, Reactogenicity and Safety of 1 Dose of GSK Biologicals' Meningococcal Vaccine GSK134612 vs. 1 Dose of Sanofi-Pasteur's Menactra® in Healthy Subjects 10-25 Years.
Brief Title: Immunogenicity and Safety of Meningococcal Vaccine GSK134612 vs. Menactra® in Healthy Adolescent/Adults Aged 10-25 Years.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 109377
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2017-04

CONDITIONS: Infections, Meningococcal
Keywords: Meningococcal Serogroups A, C, W-135 and/or Y Disease
MeSH Terms: conditions — Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Group A (Experimental): Subjects aged 10 years (< 11 years) vaccinated with meningococcal vaccine GSK134612.
  Interventions: Biological: Meningococcal vaccine 134612
- Group B (Experimental): Subjects aged 11 to 25 years vaccinated with meningococcal vaccine GSK134612.
  Interventions: Biological: Meningococcal vaccine 134612
- Group C (Active Comparator): Subjects aged 11 to 25 years vaccinated with Menactra®.
  Interventions: Biological: Menactra®

INTERVENTIONS:
Biological: Meningococcal vaccine 134612 — Single dose intramuscular injection.
  Arms: Group A; Group B
Biological: Menactra® — Single dose intramuscular injection.
  Arms: Group C

SUMMARY:
The purpose of the study is to characterize the safety and immunogenicity of 1 dose of GSK Biologicals' meningococcal vaccine GSK134612 as compared to Menactra® in adolescents/adults 11-25 years of age.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

The protocol posting has been updated following a protocol amendment.

DETAILED DESCRIPTION:
Subjects 11-25 years of age will be randomized to receive either the meningococcal vaccine GSK134612 or Menactra®. An additional non-randomized group of subjects aged 10 years (< 11 years of age) will be enrolled to receive meningococcal vaccine GSK134612 only (At the time the study begun, Menactra® was only licensed in the United States for individuals above 11 years of age and therefore could not be used as a control vaccine in subjects less than 11 years old).

This study will be single-blind for the subjects 11 to 25 years of age and open for the subjects 10 to < 11 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whom the investigator believes can and will comply with the requirements of the protocol.
* A male or female between, and including, 10 and 25 years of age (has not attained his/her 26th birthday) at the time of the vaccination.
* Written informed consent obtained from parents/guardian of the subject and written informed assent obtained from the subject if the subject is less than 18 years of age, or written informed consent obtained from the subject if the subject has achieved the 18th birthday.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception (including abstinence) for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within one month of the dose of vaccine(s).
* Previous vaccination with meningococcal polysaccharide or conjugate vaccine of serogroup A, C W-135, and/or Y.
* Previous vaccination with tetanus and diphtheria toxoids within the last month (i.e., Tdap, Td, and TT-containing vaccine within the last month).
* History of meningococcal disease due to serogroup A, C, W-135, or Y.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary), including human immunodeficiency virus (HIV) infection, based on medical history and physical examination (no laboratory testing is required).
* A family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Previous history of Guillain-Barré Syndrome.
* Bleeding disorders, such as hemophilia or thrombocytopenia, or subjects on anti-coagulant therapy.
* Acute disease at the time of enrollment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 873 (Actual)
Dates: Start 2007-04-23; Primary Completion 2007-10-31 (Actual); Study Completion 2008-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (9):
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Fairfield, California
  - GSK Investigational Site, Redwood City, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Waianae, Hawaii
  - GSK Investigational Site, Waipio, Hawaii

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Baxter R, Baine Y, Ensor K, Bianco V, Friedland LR, Miller JM. Immunogenicity and safety of an investigational quadrivalent meningococcal ACWY tetanus toxoid conjugate vaccine in healthy adolescents and young adults 10 to 25 years of age. Pediatr Infect Dis J. 2011 Mar;30(3):e41-8. doi: 10.1097/INF.0b013e3182054ab9. PMID 21200360
- [Background] Baxter R et al. Immunogenicity and safety of an investigational quadrivalent meningococcal ACWY tetanus toxoid conjugate vaccine in healthy adolescents and young adults: 1-year follow-up. Abstract presented at the 51st Annual Interscience Conference on Antimicrobial Agents & Chemotherapy. Chicago, US, 17-20 September 2011.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 109377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 873 subjects enrolled in the study, only 872 subjects received the vaccination course and started the study.
Groups:
- Nimenrix 11-25Y Group: Subjects, male or female, aged 11 to 25 years received one dose of Nimenrix™ vaccine administered intramuscularly in the deltoid region of the non-dominant arm.
- Menactra Group: Subjects, male or female, aged 11 to 25 years received one dose of Menactra® vaccine administered intramuscularly in the deltoid region of the non-dominant arm.
- Nimenrix 10Y Group: Subjects, male or female, aged 10 years (<11 years) of age received one dose of Nimenrix™ vaccine administered intramuscularly in the deltoid region of the non-dominant arm.
Period: Overall Study
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
Started | 587 | 197 | 88
Completed | 580 | 194 | 86
Not Completed | 7 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Migrated/moved from study area | 0 | 0 | 1
Not completed — Lost to follow-up (complete vaccination) | 5 | 3 | 1
Not completed — Others | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group | Total
Number analyzed (Participants) | 587 | 197 | 88 | 872
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.8 (2.69) | 14.7 (2.78) | 10 (0) | 14.29 (2.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274 | 101 | 51 | 426
  Male | 313 | 96 | 37 | 446
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 35 | 12 | 9 | 56
  American Indian or Alaskan Native | 49 | 21 | 9 | 79
  Asian-Central/South Asian heritage | 5 | 3 | 1 | 9
  Asian-East Asian heritage | 17 | 1 | 5 | 23
  Asian-Japanese heritage | 7 | 4 | 0 | 11
  Asian-South East Asian heritage | 40 | 14 | 8 | 62
  Native Hawaiian or other Pacific Islander | 4 | 2 | 1 | 7
  White-Arabic/North African heritage | 2 | 2 | 1 | 5
  White-Caucasian/European heritage | 290 | 95 | 34 | 419
  Unspecified | 138 | 43 | 20 | 201

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Bactericidal Assay Using Human Complement Against Neisseria Meningitides Serogroups A, C , W-135, Y (hSBA-MenA, hSBA-MenC , hSBA-MenW -135 and hSBA-Men-Y) Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:8.
Time Frame: At Day 0 (PRE)
Population: The analyses were performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available. The interval between Visit 1 (Month 0) and Visit 2 (Month 1) for inclusion in this cohort was defined as 21 to 48 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
Number analyzed (Participants) | 506 | 174 | 77
Participants
  hSBA-MenA: number analyzed (Participants) | 503 | 172 | 77
  hSBA-MenA | 49 | 13 | 5
  hSBA-MenC: number analyzed (Participants) | 506 | 174 | 75
  hSBA-MenC | 275 | 113 | 40
  hSBA-MenW-135: number analyzed (Participants) | 461 | 151 | 70
  hSBA-MenW-135 | 114 | 51 | 11
  hSBA-MenY: number analyzed (Participants) | 491 | 162 | 73
  hSBA-MenY | 269 | 94 | 31

2. Primary Outcome: Number of Subjects With Serum Bactericidal Assay Using Human Complement Against Neisseria Meningitides Serogroups A, C , W-135, Y (hSBA-MenA, hSBA-MenC, hSBA-MenW -135 and hSBA-Men-Y) Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:8.
Time Frame: At Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Menactra Group: Subjects, male or female, aged 11 to 25 years received on dose of Menactra® vaccine administered intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
Number analyzed (Participants) | 517 | 174 | 79
Participants
  hSBA-MenA: number analyzed (Participants) | 507 | 167 | 79
  hSBA-MenA | 415 | 118 | 70
  hSBA-MenC: number analyzed (Participants) | 510 | 173 | 79
  hSBA-MenC | 490 | 171 | 78
  hSBA-MenW-135: number analyzed (Participants) | 479 | 149 | 77
  hSBA-MenW-135 | 438 | 114 | 73
  hSBA-MenY: number analyzed (Participants) | 517 | 170 | 79
  hSBA-MenY | 492 | 139 | 76
Statistical Analysis 1: Comparison: Nimenrix 11-25Y Group vs Menactra Group; Evaluation of the immunogenicity induced by Nimenrix™ conjugate vaccine as compared to Menactra® vaccine in terms of percentage of subjects with serum bactericidal assay using human complement against N. meningitidis serogroup A (hSBA-MenA) antibody titers ≥ 1:8 one month after vaccination; Test type: Superiority; Difference in percentage = 11.2, 95% CI 2-sided [3.87 to 19.18]
Statistical Analysis 2: Comparison: Nimenrix 11-25Y Group vs Menactra Group; Evaluation of the immunogenicity induced by Nimenrix™ conjugate vaccine as compared to Menactra® vaccine in terms of percentage of subjects with serum bactericidal assay using human complement against N. meningitidis serogroup C (hSBA-MenC) antibody titers ≥ 1:8 one month after vaccination; Test type: Superiority; Difference in percentage = -2.77, 95% CI 2-sided [-5.08 to 0.40]
Statistical Analysis 3: Comparison: Nimenrix 11-25Y Group vs Menactra Group; Evaluation of the immunogenicity induced by Nimenrix™ conjugate vaccine as compared to Menactra® vaccine in terms of percentage of subjects with serum bactericidal assay using human complement against N. meningitidis serogroup W-135 (hSBA-MenW -135) antibody titers ≥ 1:8 one month after vaccination; Test type: Superiority; Difference in percentage = 14.93, 95% CI 2-sided [8.24 to 22.71]
Statistical Analysis 4: Comparison: Nimenrix 11-25Y Group vs Menactra Group; Evaluation of the immunogenicity induced by Nimenrix™ conjugate vaccine as compared to Menactra® vaccine in terms of percentage of subjects with serum bactericidal assay using human complement against N. meningitidis serogroup Y (hSBA-MenY) antibody titers ≥ 1:8 one month after vaccination; Test type: Superiority; Difference in percentage = 13.40, 95% CI 2-sided [7.90 to 20.10]

3. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW -135 and hSBA-Men-Y Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:4.
Time Frame: At Day 0 (PRE) and Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
Number analyzed (Participants) | 517 | 174 | 79
Participants
  hSBA-MenA, PRE: number analyzed (Participants) | 503 | 172 | 77
  hSBA-MenA, PRE | 68 | 18 | 7
  hSBA-MenA, Month 1: number analyzed (Participants) | 507 | 167 | 79
  hSBA-MenA, Month 1 | 421 | 118 | 71
  hSBA-MenC, PRE: number analyzed (Participants) | 506 | 174 | 75
  hSBA-MenC, PRE | 276 | 114 | 40
  hSBA-MenC, Month 1: number analyzed (Participants) | 510 | 173 | 79
  hSBA-MenC, Month 1 | 490 | 171 | 78
  hSBA-MenW-135, PRE: number analyzed (Participants) | 461 | 151 | 70
  hSBA-MenW-135, PRE | 118 | 51 | 11
  hSBA-MenW-135, Month 1: number analyzed (Participants) | 479 | 149 | 77
  hSBA-MenW-135, Month 1 | 441 | 117 | 73
  hSBA-MenY, PRE: number analyzed (Participants) | 491 | 162 | 73
  hSBA-MenY, PRE | 273 | 94 | 32
  hSBA-MenY, Month 1: number analyzed (Participants) | 517 | 170 | 79
  hSBA-MenY, Month 1 | 492 | 139 | 76

4. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW -135 and hSBA-Men-Y Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: At Day 0 (PRE) and Month 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
Number analyzed (Participants) | 517 | 174 | 79
Titers
  hSBA-MenA, PRE: number analyzed (Participants) | 503 | 172 | 77
  hSBA-MenA, PRE | 2.6 [2.5 to 2.8] | 2.4 [2.2 to 2.6] | 2.4 [2.1 to 2.9]
  hSBA-MenA, Month 1: number analyzed (Participants) | 507 | 167 | 79
  hSBA-MenA, Month 1 | 57.2 [48.8 to 67.0] | 36.0 [26.1 to 49.7] | 91.5 [64.0 to 130.8]
  hSBA-MenC, PRE: number analyzed (Participants) | 506 | 174 | 75
  hSBA-MenC, PRE | 12.8 [10.9 to 15.1] | 17.9 [13.5 to 23.6] | 9.7 [6.7 to 14.2]
  hSBA-MenC, Month 1: number analyzed (Participants) | 510 | 173 | 79
  hSBA-MenC, Month 1 | 506.7 [419.1 to 612.5] | 285.8 [214.7 to 380.5] | 765.9 [505.3 to 1160.9]
  hSBA-MenW-135, PRE: number analyzed (Participants) | 461 | 151 | 70
  hSBA-MenW-135, PRE | 5.7 [4.8 to 6.8] | 8.6 [6.1 to 12.1] | 4.2 [2.8 to 6.4]
  hSBA-MenW-135, Month 1: number analyzed (Participants) | 479 | 149 | 77
  hSBA-MenW-135, Month 1 | 124.2 [106.2 to 145.2] | 74.1 [51.1 to 107.5] | 153.8 [109.9 to 215.1]
  hSBA-MenY, PRE: number analyzed (Participants) | 491 | 162 | 73
  hSBA-MenY, PRE | 22.6 [18.3 to 27.8] | 27.6 [19.0 to 40.2] | 13.7 [8.0 to 23.6]
  hSBA-MenY, Month 1: number analyzed (Participants) | 517 | 170 | 79
  hSBA-MenY, Month 1 | 260.0 [225.2 to 300.2] | 110.6 [77.6 to 157.9] | 315.0 [223.6 to 443.7]

5. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) and the 8-day (Days 0-7) post-vaccination period
Population: The analyses were performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
Number analyzed (Participants) | 579 | 194 | 86
Participants
  Pain, Any, D0-3 | 317 | 105 | 48
  Pain, Grade 3, D0-3 | 9 | 2 | 0
  Redness, Any, D0-3 | 77 | 21 | 15
  Redness, Grade 3, D0-3 | 9 | 0 | 2
  Swelling, Any, D0-3 | 62 | 13 | 18
  Swelling, Grade 3, D0-3 | 11 | 1 | 3
  Pain, Any, D0-7 | 318 | 105 | 48
  Pain, Grade 3, D0-7 | 9 | 2 | 0
  Redness, Any, D0-7 | 77 | 21 | 15
  Redness, Grade 3, D0-7 | 9 | 0 | 2
  Swelling, Any, D0-7 | 63 | 13 | 18
  Swelling, Grade 3, D0-7 | 11 | 1 | 3

6. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as orally temperature equal to or above 37.5 degrees Celsius (°C)], gastrointestinal symptoms and headache. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) and the 8-day (Days 0-7) post-vaccination period
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
Number analyzed (Participants) | 579 | 194 | 86
Participants
  Fatigue, Any, D0-3 | 156 | 55 | 24
  Fatigue, Grade 3, D0-3 | 10 | 2 | 3
  Fatigue, Related, D0-3 | 139 | 49 | 21
  Fever (orally), Any, D0-3 | 34 | 11 | 6
  Fever (orally), Grade 3, D0-3 | 0 | 0 | 0
  Fever (orally), Related, D0-3 | 28 | 9 | 5
  Gastrointestinal symptoms, Any, D0-3 | 87 | 26 | 11
  Gastrointestinal symptoms, Grade 3, D0-3 | 4 | 2 | 0
  Gastrointestinal symptoms, Related, D0-3 | 74 | 22 | 9
  Headache, Any, D0-3 | 161 | 60 | 27
  Headache, Grade 3, D0-3 | 11 | 1 | 1
  Headache, Related, D0-3 | 139 | 51 | 21
  Fatigue, Any, D0-7 | 172 | 62 | 27
  Fatigue, Grade 3, D0-7 | 19 | 4 | 3
  Fatigue, Related, D0-7 | 147 | 53 | 23
  Fever (orally), Any, D0-7 | 41 | 16 | 7
  Fever (orally), Grade 3, D0-7 | 1 | 0 | 0
  Fever (orally), Related, D0-7 | 29 | 13 | 6
  Gastrointestinal symptoms, Any, D0-7 | 109 | 32 | 15
  Gastrointestinal symptoms, Grade 3, D0-7 | 8 | 3 | 2
  Gastrointestinal symptoms, Related, D0-7 | 86 | 24 | 9
  Headache, Any, D0-7 | 191 | 72 | 30
  Headache, Grade 3, D0-7 | 16 | 2 | 2
  Headache, Related, D0-7 | 157 | 57 | 24

7. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up period after vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
Number analyzed (Participants) | 587 | 197 | 88
Participants | 104 | 37 | 13

8. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 to Month 6
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
Number analyzed (Participants) | 587 | 197 | 88
Participants | 5 | 2 | 2

9. Secondary Outcome: Number of Subjects With New Onset Chronic Illness(es) (NOCI)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From Day 0 to Month 6
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
Number analyzed (Participants) | 587 | 197 | 88
Participants | 8 | 2 | 1

10. Secondary Outcome: Number of Subjects Reporting Rash
Description: Rash assessed was hives, idiopathic thrombocytopenic purpura, petechiae.
Time Frame: From Day 0 to Month 6
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
Number analyzed (Participants) | 587 | 197 | 88
Participants | 14 | 3 | 2

11. Secondary Outcome: Number of Subjects Reporting Adverse Events Resulting in Emergency Room (ER) Visits
Time Frame: From Day 0 to Month 6
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
Number analyzed (Participants) | 587 | 197 | 88
Participants | 24 | 9 | 2

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 4-day and 8-day post-vaccination period (Days 0-3 and Days 0-7), Unsolicited AEs: during the 31-day post-vaccination (Days 0-30), SAEs: during the entire study period (Day 0 - Month 6).
Description: The solicited local and general symptoms were collected only from those subjects who filled in their symptom sheets.
Arm/Group | Nimenrix 11-25Y Group | Menactra Group | Nimenrix 10Y Group
All-Cause Mortality (participants affected / at risk) | 0/587 | 0/197 | 0/88
Serious Adverse Events (participants affected / at risk) | 5/587 | 2/197 | 2/88
Other Adverse Events (participants affected / at risk) | 438/587 | 142/197 | 68/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix 11-25Y Group (N=587) | Menactra Group (N=197) | Nimenrix 10Y Group (N=88)
Appendicitis (Infections and infestations) | 2 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Swelling (General disorders) | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nimenrix 11-25Y Group (N=587) | Menactra Group (N=197) | Nimenrix 10Y Group (N=88)
Pain (Days 0-3) (General disorders) | 317/579 | 105/194 | 48/86
Redness (Days 0-3) (General disorders) | 77/579 | 21/194 | 15/86
Swelling (Days 0-3) (General disorders) | 62/579 | 13/194 | 18/86
Pain (Days 0-7) (General disorders) | 318/579 | 105/194 | 48/86
Redness (Days 0-7) (General disorders) | 77/579 | 21/194 | 15/86
Swelling (Days 0-7) (General disorders) | 63/579 | 13/194 | 18/86
Fatigue (Days 0-3) (General disorders) | 156/579 | 55/194 | 24/86
Fever/Orally (Days 0-3) (General disorders) | 34/579 | 11/194 | 6/86
Gastrointestinal (Days 0-3) (General disorders) | 87/579 | 26/194 | 11/86
Headache (Days 0-3) (General disorders) | 161/579 | 60/194 | 27/86
Fatigue (Days 0-7) (General disorders) | 172/579 | 62/194 | 27/86
Fever/Orally (Days 0-7) (General disorders) | 41/579 | 16/194 | 7/86
Gastrointestinal (Days 0-7) (General disorders) | 109/579 | 32/194 | 15/86
Headache (Days 0-7) (General disorders) | 191/579 | 72/194 | 30/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.